CLINICAL TRIAL: NCT03403049
Title: A Prospective Phase I Clinical Trial of Carbon Ion Radiation Therapy for Locally Advanced, Unresectable Pancreatic Cancer
Brief Title: Carbon Ion Radiation Therapy for Locally Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: Shanghai Proton and Heavy Ion Center (Other)
Responsible Party: Principal Investigator, Nitin Ohri, Associate Professor, Albert Einstein College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-5026; 261201500022C-0-0-1 (NIH)
Record Dates: First submitted 2016-03-08; First posted 2018-01-18 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Pancreatic Cancer; Cancer
Keywords: pancreatic cancer; pancreas; cancer; locally advanced; unresectable; radiation; radiation therapy; radiotherapy; carbon; carbon ion; ion
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms | interventions — Gemcitabine; Cisplatin; Capecitabine; Erlotinib Hydrochloride; Photons

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental): Dose-escalation phase I clinical study. In the initial dose levels, 'dose-escalation' refers to an increase in the radiotherapy dose delivered using carbon ion radiotherapy along with a corresponding decrease in the dose delivered using photons.
  Interventions: Radiation: Carbon Ion; Drug: Gemcitabine + Cisplatin; Drug: Gemcitabine + Capecitabine; Drug: Gemcitabine + Erlotinib; Drug: Gemcitabine; Radiation: Photon

INTERVENTIONS:
Radiation: Carbon Ion — Study subjects will receive carbon ion radiotherapy (CIRT), with daily fraction sizes of 3 GyE. The total CIRT dose will increase with each dose level. Subjects in dose level 1 and 2 will receive photon radiotherapy as well.
Drug: Gemcitabine + Cisplatin — Combined chemotherapy regimen before/after radiotherapy: gemcitabine-based chemotherapy regimen.
  All patients will have received 2-4 cycles of gemcitabine-based chemotherapy prior to study registration, with post-chemotherapy imaging demonstrating locally-advanced disease without evidence of distant metastatic disease spread. Patients who received chemotherapy regimens other than those listed above may be considered for study enrollment at the discretion of the lead investigators, provided that all other eligibility criteria are satisfied. Gemcitabine-based chemotherapy will be continued starting 3-5 weeks after completion of radiotherapy until disease progression, intolerability, or the patient's decline of chemotherapy.
Drug: Gemcitabine + Capecitabine — Combined chemotherapy regimen before/after radiotherapy: gemcitabine-based chemotherapy regimen.
  All patients will have received 2-4 cycles of gemcitabine-based chemotherapy prior to study registration, with post-chemotherapy imaging demonstrating locally-advanced disease without evidence of distant metastatic disease spread. Patients who received chemotherapy regimens other than those listed above may be considered for study enrollment at the discretion of the lead investigators, provided that all other eligibility criteria are satisfied. Gemcitabine-based chemotherapy will be continued starting 3-5 weeks after completion of radiotherapy until disease progression, intolerability, or the patient's decline of chemotherapy.
Drug: Gemcitabine + Erlotinib — Combined chemotherapy regimen before/after radiotherapy: gemcitabine-based chemotherapy regimen.
  All patients will have received 2-4 cycles of gemcitabine-based chemotherapy prior to study registration, with post-chemotherapy imaging demonstrating locally-advanced disease without evidence of distant metastatic disease spread. Patients who received chemotherapy regimens other than those listed above may be considered for study enrollment at the discretion of the lead investigators, provided that all other eligibility criteria are satisfied. Gemcitabine-based chemotherapy will be continued starting 3-5 weeks after completion of radiotherapy until disease progression, intolerability, or the patient's decline of chemotherapy.
Drug: Gemcitabine — Combined chemotherapy regimen before/after radiotherapy: gemcitabine-based chemotherapy regimen.
  All patients will have received 2-4 cycles of gemcitabine-based chemotherapy prior to study registration, with post-chemotherapy imaging demonstrating locally-advanced disease without evidence of distant metastatic disease spread. Patients who received chemotherapy regimens other than those listed above may be considered for study enrollment at the discretion of the lead investigators, provided that all other eligibility criteria are satisfied. Gemcitabine-based chemotherapy will be continued starting 3-5 weeks after completion of radiotherapy until disease progression, intolerability, or the patient's decline of chemotherapy.
Radiation: Photon — During this study, the prescribed dose shall be administered according to the dose escalation shown in the table, starting with dose level 1. The carbon ion dose shall be gradually escalated while gradually reducing the dose of photons until eventually administering a full dose of 56 GyE/14 Fx carbon ions (fractional dose of 4 GyE). Dose escalation will be performed in parallel for two patient groups: patients whose pancreatic tumors are greater than 5 mm from the duodenum (Group A) and those whose tumors are within 5 mm of the duodenum (Group B). Enrolled patients will be monitored for 90 days after radiotherapy starts for any acute toxic reaction and to explore the maximum tolerated dose, in addition to being observed for any related long-term toxic reactions in accordance with the protocol.

SUMMARY:
This is a phase I trial to determine the maximum tolerated dose of carbon ion radiotherapy for the treatment of locally advanced, unresectable, pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Signed the informed consent form;
2. Age ≥ 18;
3. Capable of following the protocol
4. Cytologically or histologically proven diagnosis of adenocarcinoma of the pancreas;
5. Unresectable adenocarcinoma of the pancreas by radiographic criteria according to the criteria of the NCCN Guidelines and based on post-chemotherapy imaging or due to medical contraindications to radical resection;
6. No evidence of distant metastases based on imaging evaluation;
7. Maximum tumor and positive lymph node diameter ≤ 6 cm;
8. ECOG Performance Status 0-1;
9. Life expectancy ≥ 12 weeks;
10. Adequate blood function: absolute neutrophil count (ANC) ≥1.5 x 109/L, platelet count ≥100 x 109/L, and hemoglobin ≥9 g/dL (use of transfusion to achieve said levels or greater is acceptable);
11. Adequate liver function: total bilirubin <1.5 x ULN, and AST and ALT <2.5 x ULN;
12. Adequate kidney function: serum creatinine ≤1.25 x ULN or calculated creatinine clearance rate ≥50mL/min and urine protein <2+.If the patient's baseline urine protein is at ≥2+, urine samples must be taken for 24 hours to verify that urine protein is ≤1g;
13. Laboratory studies within 14 days prior to registration demonstrating that the internationalization standard ratio (INR) ≤1.5 and prothrombin time (PPT) ≤1.5 x ULN.
14. Prior receipt of 2-4 cycles of Gemcitabine-based systemic chemotherapy.

Exclusion Criteria:

1. Lack of pathologic confirmation of pancreatic malignancy prior to treatment initiation;
2. ECOG Performance Status >=2;
3. Poor liver, kidney and bone marrow function that do not meet the requirements for treatment;
4. Persistent grade ≥ 2 toxicity due to previous cancer treatment;
5. Patient has previously received abdominal radiation therapy or abdominal radioactive seed implantation;
6. Those wearing a cardiac pacemaker or another type of metal prosthetic implant whose normal functions may suffer interference from high energy radiation or that could affect the radiation target area;
7. Where it is not possible to achieve the predetermined safety dose limit with the dose equivalent limit of the organ at risk such as the liver or digestive tract, etc.;
8. If the doctor determines that the heavy proton or carbon ion dosage radiotherapy will not bring any benefit to the patient;
9. Patients suffering from another illness or other factors that could affect the proton or carbon ion therapy;
10. Pregnant (verified by serum or urine β-HCG test) or breastfeeding females;
11. Drug-abuse or alcohol dependency;
12. HIV positive, including those that have received antiretroviral therapy; replicative stage of chronic Hepatitis B virus; active stage of Hepatitis C; and active stage of syphilis;
13. HBV positive patients suffering from replicative stage of hepatitis virus, requiring antiretroviral therapy but cannot due to a concomitant disease;
14. Patients with a history of mental illness that may prevent their completion of treatment;
15. Patients with serious complications that could affect the course of treatment, including:

    * Unstable angina, congestive heart failure, or myocardial infarction requiring hospital admittance over the last 6 months;
    * Acute or systemic bacterial infection;
    * Chronic exacerbated obstructive pulmonary disease or other respiratory system disease requiring inpatient treatment;
    * Impaired liver function or impaired kidney function;
    * Patients suffering from immunosuppression;
16. Patients with contraindications to receiving radiotherapy, such as a serious connective tissue disease (eg: scleroderma)
17. Patients that are unable to understand the objective of the treatment/cannot sign the informed consent form;
18. Patients that lack civil capacity to act or whose civil capacity to act is limited.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2019-07-09 (Actual); Study Completion 2019-07-09 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity | 90 days
  Any CTCAE v. 4.03 non-hematologic adverse event of grade 3 or higher or any hematologic adverse event of grade 4 or higher, occurring within 90 days of the start of radiotherapy and deemed to be related to carbon ion radiotherapy.

SECONDARY OUTCOMES:
Any grade 2 or higher treatment-related toxicity, scored using CTCAE v. 4.0 | through study completion, an average of 1 year
  Any grade 2 or higher treatment-related toxicity, scored using CTCAE v. 4.0
Radiographic changes following completion of study therapy (RECIST v. 1.1) | through study completion, an average of 1 year
  Radiographic changes following completion of study therapy (RECIST v. 1.1)
Overall survival duration | through study completion, an average of 1 year
  The length of time from study inclusion until death from any cause
Progression-free survival duration | through study completion, an average of 1 year
  The length of time from study inclusion until death from any cause or disease progression at any site
The impact in terms of overall quality of life of radiation therapy as assessed by the QLQ-C30 questionnaire | through study completion, an average of 1 year
  Quality of life will be assessed at various time points using the European Organisation for Research and Treatment of Cancer 30 items dealing with fatigue, pain, nausea and vomiting, general condition and social, emotional and cognitive functions. It is currently used in many cancer related clinical trials.

CONTACTS AND LOCATIONS:
Overall Officials: Chandan Guha, M.B.B.S., Ph.D., Principal Investigator — Albert Einstein College of Medicine
Locations (2):
- Albert Einstein College of Medicine, The Bronx, New York, United States
- Shanghai Proton and Heavy Ion Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided